CLINICAL TRIAL: NCT06459544
Title: Effects of Bobath Approach With Core Stability to Improve Balance in Stroke
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: MSRSW/Batch-Fall22/726
Record Dates: First submitted 2024-06-10; First posted 2024-06-14 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Balance; Distorted
MeSH Terms: interventions — Core Stability

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bobath Technique with core stability (Experimental)
  Interventions: Diagnostic Test: Bobath Technique with core stability
- Conventional treatment for balance (Other)
  Interventions: Other: Conventional treatment for balance

INTERVENTIONS:
Diagnostic Test: Bobath Technique with core stability — exercise to improve balance motor learning stretegy is basically used. Bobath in which we assess patient's posture, inhibit the abnormal muscle tone and facilitate normal patterns and posture through handling and posture. we also use sensory inputs like propioception to promote normal pattern. we take some exercise based on bobath technique with core stability like Bridging with core stability, quadroped with core stability, sitting and standing with core stablity, single leg standing , dynamic balance with core stability.treatment plan based on 45 minutes per day, 6 days a week for 4 week.
  Arms: Bobath Technique with core stability
Other: Conventional treatment for balance — like stretching, strenthening the Lower extremity muscles , PROMS, AAROMS,AROMS, RROMS,some balance exercise like sitting and standing
  Arms: Conventional treatment for balance

SUMMARY:
Bobath technique with core stability exercises to improve balance in stroke. Randomized clinical trial study design will be followed. Data will be collected from following centers: Naseer Hospital, North Ravi Hospital, Bajwa Hoaspital,Minhaj Physiotherapy Centre, Home visits. Probability Random Sampling is used.

ELIGIBILITY:
Inclusion Criteria:

* age 30 - 65
* Both Gender
* more than 1 month or less than 6 months since onset of stroke
* GCS SCORE 11 TO 15

Exclusion Criteria:

* consist of GCS less than 10
* any pathological fracture
* diagnosed orthostatic hypotension
* Comorbidities like IHD and Rheumatologic disease.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-10-30 (Estimated)

PRIMARY OUTCOMES:
Balance berg scale | 12 Months
  Evaluates balance during a sequence of pre-planned tasks in an objective manner. It takes 20 minutes and consists of 14 tests. It is 5 points ordinal scale with 0 = lowest degree of function and 4 = highest level. The highest score is 14
Trunk Impairment Scale | 12 months
  Evaluate static and dynamic balance and trunk coordination.score goes from 0 = lowest performance and 23 = highest performance. Scores vary from 0 to 16.

CONTACTS AND LOCATIONS:
Locations (1):
- Naseer Hospital 16 A , AHMAD BLOCK NEW GARDEN TOWN, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No